CLINICAL TRIAL: NCT06871488
Title: Identification of Neural Markers of Aggression and Irritability and Their Capacity to Predict Treatment Response to CNS Stimulant Medication in Youth With ADHD
Brief Title: Predictors of Improvements in Irritability and Aggression in Children With ADHD Treated With CNS Stimulants
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, James Waxmonsky, Professor of Psychiatry, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MH137647
Record Dates: First submitted 2025-02-14; First posted 2025-03-12 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: ADHD - Attention Deficit Disorder With Hyperactivity; Irritability; Aggression Childhood
Keywords: ADHD; CNS Stimulants; Irritability; Aggression
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Aggression | interventions — Central Nervous System Stimulants; Clinical Trials, Phase II as Topic

STUDY DESIGN:
Intervention Model Description: two phases- first is single group open label to identify optimal dose followed by blinded randomized within subjects crossover design of optimal dose vs placebo for each participant
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: the child participants primary school teacher (secondary outcomes assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Blinded optimal dose (phase two) (Active Comparator): In this second treatment phase of the study, all participants will receive under blinded conditions their optimal dose of CNS stimulant from the prior phase for a total of 7 days
  Interventions: Drug: CNS Stimulant
- Placebo (phase two) (Placebo Comparator): In this second treatment phase of the study, all participants will receive placebo under blinded conditions for a total of 7 days
  Interventions: Drug: Placebo
- open label dose optimization (phase one) (Experimental): In this first treatment phase, all participants will have their dose of CNS Stimulant optimized over 6 visits under open label conditions. This arm will use any FDA approved CNS stimulant for pediatric ADHD at their approved dose. By the end of this phase, the optimal dose for the next phase will be identified.
  Interventions: Other: CNS Stimulant open label first phase

INTERVENTIONS:
Drug: CNS Stimulant — The second treatment phase (blinded within subjects crossover) will compare one week of the optimal dose of CNS Stimulant (from the prior phase) to one week of placebo for a total of 14 days of data collection.
  Other Names: CNS Simulant RCT phase (second phase)
  Arms: Blinded optimal dose (phase two)
Drug: Placebo — Placebo is only used during the second of two treatment phases. The second treatment phase (blinded within subjects crossover) will compare one week of the optimal dose of CNS Stimulant (from the prior phase) to one week of placebo.
  Arms: Placebo (phase two)
Other: CNS Stimulant open label first phase — The first treatment phase will optimize CNS stimulant dose under open label conditions using any approved FDA medication for pediatric ADHD at the FDA approved doses.
  Arms: open label dose optimization (phase one)

SUMMARY:
Impulsive Aggression and chronic irritability (IACI) often occur together and are one of the most common reasons children present for behavioral health (BH) care. ADHD frequently associated with IACI as upwards of 50% of youth with ADHD manifest impairing IACI levels. IACI is the most common reason that children with ADHD are prescribed antipsychotics and admitted to inpatient BH units. Systematic dose optimization of CNS stimulants improves levels of IACI, reducing the need for these more intensive and burdensome treatments. However, response varies, with over half of children with ADHD showing meaningful improvement, upwards of 40% receiving minimal benefit and 3 to 10% exhibiting increased IACI levels. Symptom levels of ADHD or IACI and other demographic variables are of limited utility for predicting response, suggesting the need to move beyond symptoms in the search for treatment predictors. Youth with ADHD and IACI struggle with multiple aspects reinforcement learning (RL), defined as learning from interactions with the environment to reach a goal. Successful RL efforts tap multiple cognitive functions. In controlled laboratory tasks, youth with IACI and various BH disorders exhibit excessive behavioral and neural response to receiving reward (reward responsiveness), difficulty processing environmental cues to adapt behavior to meet a goal (set shifting/goal updating) and impaired ability to flexibly attend to relevant stimuli when blocked from a goal (frustrative nonreward). Event related potentials (ERP) are small electrical responses in the brain in response to specific events or stimuli measured by electroencephalogram (EEG) testing. ERPs exist that can serve as established neural measures of each of these cognitive functions offering a child friendly means to assess their contribution to observable levels of IACI.

CNS stimulants improve functioning in these specific realms and impact associated ERPs to the degree that differences between ADHD and non-ADHD youth disappear. This study will examine the capacity of these ERPs to predict levels of IACI exhibited by children with ADHD when at home. Investigators will then assess if variability across children in the capacity of CNS stimulants to impact RL associated ERPs accounts for differences in the clinical effects of CNS stimulant medications to improve IACI at home using a multimethod battery integrating ERPs, parent report and task performance. Specifically, investigators will examine variance in the reward positivity (RewP) ERP when receiving reward feedback, the switch positivity (SwP) ERP measuring mental effort when cued to shift set and the change in P3b amplitude measuring attention allocation when transitioning from reward to nonreward on a go-no-go task. To achieve these aims, 136 children with ADHD and elevated IACI levels will have their CNS stimulant dose optimized over six weeks and then complete a two week within subjects crossover trial of placebo versus optimal dose. ERP collection will be completed within each blinded week. Parent ratings will be gathered 3 times per day including during peak and off-peak times of medication efficacy to capture the variance in IACI levels within the day and disentangle reports of worsening IACI related to loss of previously beneficial medication effects versus those most likely related to a direct adverse response to medication.

DETAILED DESCRIPTION:
This is clinical trial of CNS stimulants will enroll 136 youth with ADHD and elevated levels of impulsive aggression and chronic irritability (IACI). It employs a 6 week open label dose optimization trial followed by a 2 week within subjects crossover phase of optimal dose versus placebo. In our preliminary work, the study team observed that about 50 to 60% of children will show moderate or greater improvements in IACI with CNS Stimulants dose optimization. This response appears independent of ADHD symptom change. Across studies, 5 to 10% of youth with ADHD experience increased IACI, but there are no reliable predictors of IACI worsening. Youth with IACI have multiple impairments with reinforcement learning that can manifest at the neural level as altered event response potentials (ERP) and at the behavioral level as impaired cognitive task performance. For example, investigators demonstrated that youth with IACI showed enhanced response to reward feedback and reduced capacity to allocate attention under frustration manifesting as alterations in the amplitude of the Reward Positivity (RewP) and P3b ERPs respectively. Others have demonstrated that youth with IACI have impairments in shifting set as captured by the switch positivity ERP (SwP). Not such impairments are seen in youth with ADHD but not elevated IACI levels. All three of these ERPs are impacted by CNS stimulants, and these medications have been shown to improve reinforcement learning (RL) in youth with ADHD when it is impaired. Therefore, the study team theorizes that the degree of IACI improvement in IACI seen with CNS stimulants will correlate with the level of ERP amplitude change seen with these medications.

To test this theory, investigators will recruit 136 youth ages 8 to 12 with ADHD and elevated levels of IACI. All participants will first have their stimulant dose optimized (any oral FDA approved stimulant for ADHD that be can blinded) over 6 weekly visits using weekly ratings gathered from guardians and teachers. If ADHD symptoms show a 25% or greater improvement and there is not a moderate worsening in IACI levels (it is expected that 50%or more of participants will show reduced levels, 35% little change, 5-10% mild worsening and few if any will show moderate or worse impairment), then participants will be advanced to a 2 week within subjects double blind randomized controlled trial (RCT) phase using a within subjects crossover design with each participant receiving their optimal dose of CNS stimulant and placebo for one week apiece. A thrice daily ecological momentary assessment (EMA) protocol measuring ADHD and IACI levels will be completed in each of these two weeks levels to address the appreciable temporal fluctuations in IACI seen across the day at home. In each blinded week, guardians will complete three ratings per day of IACI and ADHD. During times when medication effects are active, participants will complete an approximately one-hour EEG testing battery within each condition (once on med/ once on placebo) measuring these ERP amplitudes. Participants, guardians and study staff will be masked to intervention status during the RCT phase but not the open label dose optimization phase. All EEG data collection will occur under blinded conditions. This within subjects design reduces inter subject variance which is essential for identification of treatment biomarkers by predetermining each participants optimal dose and then using each participant as their own control.

Participants will be 136 youth with ADHD and elevated levels of IACI ages 8 to 12. Elevated levels of IACI will be defined by guardian rating on the Affective Reactivity Index (ARI) and Revised Modified Overt Aggression Score (RMOAS) as both are representative of an impairing level of IACI. Children will also be required to have at least moderate impairment (4+) on the Impairment Rating Scale (IRS) and the ADHD Clinical Global Impressions Severity Score (CGI-S) and meet full diagnostic criteria for ADHD. ADHD will be assessed using the Disruptive Behaviors Disorder Guardian Interview given by masters level staff. It assesses all ADHD symptoms and all other DSM ADHD criteria. The guardian interview will be supplemented with teacher ratings of ADHD (Disruptive Behavior Disorder Rating Scale [DBD-RS]) and classroom functioning (IRS) to verify impairment and symptoms occur across settings. A dual clinician review by study MD/PhD will make a final diagnosis by integrating teacher and guardian report using the OR rule. Where disagreement occurs, a third clinician will be consulted. Many youth with ADHD and elevated IACI have comorbid behavioral health conditions. Consistent with past ADHD trials for IACI, investigators will exclude youth with prominent autism traits (defined as mean score above 3.2 on the Autism Symptoms Dimension Questionnaire) or current major depression. However, anxious or subthreshold depressive symptoms do not impede the ability of CNS stimulants to improve ADHD or IACI. Comorbid conditions will be assessed on the Kidde Schedule for Affective Disorders and Schizophrenia Computerized Version (KSADS-Comp). To better examine their impact on planned outcomes, depression and anxiety symptoms will also be measured dimensionally by guardian and youth report on the Revised Children's Anxiety and Depression Scale-25 (RCADS-25). Stimulant optimization is advised before considering other psychotropics for aggression, so antipsychotics will be exclusionary. Antidepressants, alpha agonists and psychotherapy will be allowed and examined as covariates if dose has been stable for 30+ days as they do not meaningfully change amplitude of the selected ERPs or the response to CNS stimulants. Doses of outside medication and therapy frequency/format/modality must be held stable for study duration. Children who lack the cognitive, visual or auditory capacity to complete laboratory tasks or have a medical/psychiatric contraindication to CNS stimulants will be excluded as will youth with 2+ fully optimized methylphenidate trials AND 2+ amphetamine trials. This last requirement should not lead to appreciable exclusions as CNS stimulants are often not titrated to optimal doses. Youth who are stimulant naïve will be allowed to enroll as long as they meet enrollment criteria and do not have medical conditions that would preclude use of CNS stimulants (seizure disorder, significant structural cardiac abnormalities, severe tics, etc.). Study staff will meet with families to review study goals and commitments and complete consent and assent. During the intake assessment, a MD clinician will complete a thorough medication history to review past medication trials of CNS stimulants as well as health variables that may impact tolerability of CNS stimulants (e.g. sleep and appetite). The clinician driven ADHD RS 5 interview and the clinician driven ARI interview (C-ARI) will be completed to assess current level of ADHD symptoms and IACI levels and repeatedly weekly during the dose optimization phase. The Clinician-ARI Interview is a semi structured interview which codes levels of IACI on a 0-100 metric with separate ratings for levels of irritability and aggression, based on ratings of frequency, duration and severity for each. This relatively new measure will provide critical information about the timing of IACI, assisting with medication selection. It will be repeated at the end of dose optimization phase as part of a multimethod battery of IACI to compare agreement between guardian ratings of IACI and clinician assessment.

Dose Optimization Phase: An initial medication option will be selected based on the participant's past medication trials and current temporal patterns of impairment (time of day of greatest impairment) with a focus on improving ADHD levels across the day and IACI levels at home. All study medication will be prescribed by licensed physicians expert in the treatment of pediatric ADHD and IACI (three child psychiatrists and one general pediatrician that are study investigators). All study treatments consist of only CNS stimulants approved for the treatment of pediatric ADHD or placebo. Methylphenidate will be the preferred initial option based on prior IACI treatment trials but amphetamine products will also be allowed; however, any FDA approved medication in either of these stimulant classes can be employed as long as it can be blinded for the RCT phase (no liquids or dissolve tabs or transdermals unless our research pharmacy can obtain a comparable blind). Children will be taught to swallow capsules during the open label medication phase using established procedures from past trials in this same population. The employed dosing will be consistent with standard clinical practice and past trials in youth with IACI and ADHD, with doses adjusted by one dosing increment at a time. During the 6 week dose optimization period, study clinicians will adjust dose using weekly guardian and teacher ratings collected and direct interview of guardian using the ADHD RS 5 interview until optimal dose is achieved based on efficacy and tolerability ratings. Participants will complete weekly visits with study physicians to adjust CNS stimulant dose. At each weekly visit, guardians will complete the ARI and R-MOAS, a brief measure of functional impairment (IRS) as well medication tolerability with the Pittsburgh Side Effect Rating Scale (PSERS). Guardians will also be asked to identify for each dosing the day, the hour when medication benefits appear to onset and the hour when they appear to have fully dissipated in order to identify medicated and unmedicated time periods of the day to be used to define the EMA sampling times for the following RCT stage. Clinicians will complete the ADHD-RS interview to measure change in ADHD symptoms and the Clinical Global Impressions Severity and Improvement Scale (CGI S and I) separately for ADHD and IACI to assess change in each since baseline and total current severity of each construct over the past week. Every week, teachers will be sent a link to a secure survey for them to rate the current level of ADHD symptoms and oppositional behaviors (IOWA Conners) and IACI levels at school (6 item teacher version of ARI and 6 item abridged RMOAS). Clinicians will also complete the Columbia Suicide Severity Rating Scale (C-SSRS) each week with participants and guardians to measure risk for self-harm. In addition, guardian ratings of Oppositional Defiant Disorder and Conduct Disorder (DBD-RS will be collected). Expanded teacher ratings of ADHD, Conduct Disorder and Oppositional Defiant Disorder that capture every DSM symptom will also be collected at endpoint (DBD RS). Vitals (height, weight, blood pressure, pulse) will be collected at every in person office visit, with in-office visits required at least every two weeks. Alternating visits can be done via HIPAA compliant telehealth platforms. The dose optimization period can last up to 6 weeks but may end sooner if participants meet criteria for optimal dose. For dose to be considered optimal and the titration to end before week 6, CGI improvement (CGI-I) ratings for ADHD must be at much be much or very much improved levels with acceptable medication tolerability for at least two consecutive visits with clinicians deeming that further improvement is not expected or higher doses could not be tolerated. The study team has employed this same definition in prior NIH studies (MH083692). Once dose has been optimized, participants will be advanced to the next phase. As this study aims to identify markers of CNS stimulant response for IACI, it is important to assess predictors in participants evidencing a wide range of responses for IACI when treated with CNS stimulants versus limiting biomarker assessment to only robust responders. However, study treatments will only be continued in those participants evidencing at least partial improvement in ADHD symptoms (the FDA approved indication for all study medications) to ensure that all participants advancing to the next phase are experiencing some benefit. Similar criteria were used in past adjunctive pharmacotherapy trials for IACI. The ADHDRS-5 will be employed as the primary gating measure to ensure participants meet response criteria to advance to the next phase as study medications are FDA approved for treatment of ADHD versus IACI. Consistent with past ADHD trials, the threshold for ADHD response will be defined as at least a 25% improvement in ADHD symptoms as measured by the ADHD RS. To advance to the next stage, participants must also display improved, comparable or mildly worse IACI levels (any option except "much" or "very much" worse on IACI CGI-S). Based on prior work it is expected that 80% or more of youth will meet criteria to advance to the randomized controlled (RCT) phase.

RCT phase: Once participants complete the open label phase, they will be randomly assigned in a balanced fashion to one of two medication sequences (medication - placebo or placebo-medication). Dropout for other reasons or data loss is not estimated to be more than 10%, leaving at least 96 participants with full study data. The RCT phase will consist of two randomly assigned 7 days stretches of blinded optimal dose or matching placebo beginning on a Saturday and ending on a Friday. The order will be randomly assigned across participants (medication - placebo vs placebo-medication). An EEG testing battery will be completed once per week in each arm at a time when medication has been deemed to be active consistent with the extant literature and guardian report of medication effects during the open label dose optimization.

The guardian and child will also come to the clinic for a weekly medication visit to assess medication tolerability, collect vitals and complete clinician ratings (see below). If the testing visit occurs early in the blinded week limiting the duration of assessment, then vitals will be collected and guardians and clinician will complete a telehealth med visit later in the week to complete guardian and clinician driven measures. Treatments will be blinded to the study team, guardian and participant during the two week within subject's crossover phase. This design is commonly used in FDA approval trials of new CNS stimulants for pediatric ADHD with little evidence of crossover effects or guessing the blind. The Penn State College of Medicine Investigational Drug Service will prepare blinded capsules for this study. The active capsules will consist of the tablet or capsule of the commercially available medication being placed in a gelatin capsule with a filler such as methylcellulose. Placebo capsules will consist of a gelatin capsule filled with a filler such as methylcellulose. The same size and color of gelatin capsule will be used to prepare both the active and placebo capsules so that all but the pharmacists remains blinded. Any pill products will be encapsulated with participants trained to swallow capsules during the 6 week open label using procedures successfully employed in our past trials. Participants and their families will be dispensed one week of placebo or blinded medication at a time in a labeled pill blister packet to reduce chances of dosing error. Dosing prompts will be sent out each morning and guardians will be asked to report time of dosing in the EMA survey. Pill counts will also be completed at each visit in this phase. The investigational drug service will hold the blind which can be broken 24 hours per day by contacting the pharmacist on call if a serious adverse event arises. Guardians will complete an ecological momentary assessment (EMA) battery 3x per day for 7 days (Saturday to Friday), rating CI on the first six items of the ARI. For IA, the study team will use a 6-item abridged version of the R-MOAS with 2 items each from the verbal aggression, physical aggression and aggression to property subscales. At each time, guardians will also rate ADHD symptoms on the 5 item IOWA Abbreviated Conners, time spent with the child that period (if <15 mins, survey ends) and settings where they interacted (home, school, structured extracurricular, unstructured peer interaction, out of house with family). Daily, they will rate when study medication was taken, if medication onset and offset was as expected (based on titration phase) and the time taken to fall asleep, time awake once first falling asleep and time awake in morning as these items correlate with IACI levels. The study team will employ event-based sampling centered around perceived timing of medication effects. Each day, guardians will be asked to rate the child's behavior before the study med is perceived to be active (T1: typically first 1-2 hours of day), the time medication appears active at home (T2) (afternoon into early evening) and the time from when med appears to have worn off until the child is asleep (T3:typically last 1-2 hours of day). Even with extended release preps, guardians can detect medicated and unmedicated times in the evening. The exact times for each assessment period will be established during the open label phase based on observed onset and offset of the optimized stimulant dose. Sampling times can be adjusted across days to account for differences in med administration on school and non-school days. Survey data will be collected via the LifeData application which alerts guardians when a survey is due and then transmits all collected data to a secure server. A study staff member will download a survey application directly to the family's smart phone as well as instructions on how to complete the EMA surveys. The survey application will signal them after the preselected times to complete a rating. All data is encrypted on the phone and transmitted directly to a secured server. Prior work has found that guardians will complete over 85% of EMA ratings in a 30-day period. Our lab has employed similar surveys of guardians with over comparable completion rates (see prelim studies). If this completion rate is achieved, then 18 ratings will be captured per week. The combined measures can be completed in under 10 minutes as they total no more than 30 questions. Each week, teachers will also be asked to complete a weekly rating of IACI (Teacher rated ARI/abridged RMOAS) and ADHD symptoms (IOWA). Each week, guardians will also complete the PSERS and IRS. Weekly, clinicians will complete the CGIs and C-ARI interview with guardians to comprise a multimethod assessment of IACI over the entire week. Once this phase is done, participants and guardians will attend a final close out visit to review results and plan for aftercare, with ongoing specialty behavioral health care offered in Penn State Psychiatry.

EEG Assessment: Participants will complete an identical battery of cognitive tasks assessing reinforcement learning capacity under EEG collection in each of the two blinded RCT weeks at a time when medication has been deemed active based on the prior dose of the optimization phase and the extant psychopharmacology literature. This battery will measure the selected ERPs associated with reinforcement learning (RL). The frustrative non-reward task will always be done last to prevent carryover effects from emotional arousal to the other two tasks, whose order will be randomized across visits (set shifting versus simple guessing task). All testing will be completed at the Penn State Health Ambulatory EEG lab which is located directly in the primary outpatient behavioral health clinic, which is the main referral site for the study. It is also the location for the Penn State Health Attention and Behavior Clinic where all other study visits will occur. All ERP assessments will take place with the child seated at a table with a computer monitor and keyboard (or response box). One research assistant is stationed next to the child and the second is beyond the child monitoring data collection. Cap size will be selected based on participant's head circumference and placed according to anatomical standards. Three different aspects of reinforcement learning will be assessed at this session: reward responsiveness, set shifting and attentional allocation under reward and nonreward.

Reward Responsiveness: The experimental task used to elicit event-related potentials to reward and loss feedback will be a simple guessing reward task shown in previous research to reliably elicit the reward positivity ERP (RewP) in children and adolescentsThe primary analysis for this task will be change in amplitude for residual score between medication and placebo for RewP wins as more consistent effect of CNS stimulants has been observed for wins than losses.

Set shifting/goal updating task: This will be measured with a cued switch task using a variant of the NAVON test. A global figure (e.g. "S") comprised of smaller local letters (e.g. "H's") is presented on the monitor (Figure 6). Participants are instructed to press a button identifying the correct figure based on whether they are cued to attend to the global or local letter amongst four possible options (local icon, global icon or two icons unrelated to either letter). Regression analyses will be conducted to create residuals reflecting the difference in amplitude for the switch and stay positivity, with SwP as the dependent variable (SwP residual) to isolate changes in the ERP wave attributable to cognitive processes involved in set shifting.

Frustrative Nonreward: The goal of this task is to measure cognitive processing changes in the context of frustration versus reward to examine the impact of affect on attentional deployment as indicated by the P3b amplitude during a Go/no-go task. The study team will use comparable procedures to those employed in our prior work (see prelim studies). For the Go/no-go task, children are instructed to "zap' alien invaders by pressing a button but advised to not stop an alien that appears two times in a row. A red box appears around the visual stimulus when a mistake is made (zap a no-go stimulus or fail to zap a go). There are 3 blocks with the first favoring point accumulation by awarding more value to correct versus incorrect answers. The second is the frustration block where point assignment is reversed such that all participants will experience some degree of net loss of points designed to induce frustration. The third block uses the same scoring algorithm as the first assuring that all finish with a positive point total.

ELIGIBILITY:
Inclusion Criteria:

1. Meet criteria for any presentation of ADHD
2. Moderate or worse impairment related to ADHD
3. Elevated levels of irritability and/or aggression on guardian ratings of Affective
4. Reactivity Index and Retrospective Modified Overt Aggression Scale
5. fluent in English for child and guardian
6. Guardian and child are willing to have child take CNS stimulant medication for ADHD

Exclusion Criteria:

1. Medical contraindications to use of CNS stimulants
2. Autism Spectrum Disorder,
3. Bipolar Disorder,
4. Intellectual/Developmental Delay
5. current use of antipsychotic, mood stabilizing
6. Use of other medications that impact EEG data collection (e.g. benzodiazepenes)
7. hearing or visual deficits that impede ability to do computer tasks
8. Current Major Depressive Episode
9. Current suicidal ideation
10. child has failed two fully optimized trials of methylphenidate products AND amphetamine products

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 136 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2030-02-28 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
RCT phase: Guardian rated Affective reactivity Index (ARI) | 7 days on med and for 7 days on placebo for 14 days of data collection
  Thus study examines response markers for CNS stimulants to improve irritability and to improve aggression. For this second treatment phase comprised of the within subjects crossover of optimal med vs placebo, the primary outcome for irritability is the drug placebo difference in the guardian rated Affective Reactivity Index collected for 7 days over the blinded within subjects crossover phase. ARI has 6 items rated 0-2 for range of - to 14 with higher scores representing greater irritability levels. drug placebo difference on this measure will be correlated with drug placebo difference for RewP, P3b and switch positivity ERP
Open label dose opt: ADHD RS 5 clinician interview | 6 visits (over a max duration of 12 weeks)
  For the first treatment phase (open label dose optimization) the primary outcome is the change in ADHD symptoms as measured by clinician interview using the ADHD RS 5. it has 18 items rates 0-3 with more symptoms reflecting higher scores. will measure change over time with drug;
RCT phase abridged Revised modified overt aggression scale (RMOAS) | 7 days on med and 7 days on placebo for 14 days of data collection
  The primary rating for aggression is the drug placebo difference in the guardian rated abridged (6 reduced to 6 items) Retrospective Modified Overt Aggression Scale (RMOAS) collected for 7 days over the blinded within subjects crossover phase. The RMOAS abridged version has 6 items rated 0-3 with higher scores equating to greater levels of aggression ; drug placebo difference on this measure will be correlated with drug placebo difference for RewP, P3b and switch positivity ERP

SECONDARY OUTCOMES:
Open label dose opt: affective reactivity index -guardians (ARI) | every visit (every 1-2 weeks over max of 12 weeks)
  completed every visit in open label dose opt phase by guardians. range is 0-12 with higher scores meaning more irritability; will examine change over time with med
Open label dose opt: affective reactivity index teachers (ARI) | every visit (every 1-2 weeks over max of 12 weeks)
  completed every visit in open label dose opt phase by teachers. range is 0-12 with higher scores representing more irritability; will examine change over time with med
Open label dose opt: RMOAS by guardians | every visit (every 1-2 weeks over max of 12 weeks)
  completed at every visit in this phase by guardians ; 12 items with first 4 items having 3 item likert and next 12 having 14 item likert; weighted score 0-20 for first 4 items measuring verbal incidents, 0-120 for next 4 items measuring incidents towards others and 0 to 60 for final set of 4 items measuring incidents to property for total range of 0 to 200 with higher scores meaning more aggressive behaviors; will examine change over time with med
Open label dose opt: RMOAS by teachers | every visit (every 1-2 weeks over max of 12 weeks)
  completed at every visit in this phase by teachers; 12 items with first 4 items having 3 item likert and next 12 having 14 item likert; weighted score 0-20 for first 4 items measuring verbal incidents, 0-120 for next 4 items measuring incidents towards others and 0 to 60 for final set of 4 items measuring incidents to property for total range of 0 to 200 with higher scores meaning more aggressive behaviors; will examine change over time with med
Columbia Suicide Severity Rating Scale (CSSRS) | every visit (every 1-2 weeks over max of 12 weeks)
  completed at every visit in open label dose opt and randomized crossover phase; each item is answered yes/no and scored individually
RCT phase: Clinical Global Impressions: Impairment and Severity (CGI I/S) | weekly for 2 weeks
  completed at every visit in each of two weeks; 1 item each for impairment and severity on 1 to 7 likert; higher numbers mean more seveirty and less improvement; will examine drug placebo difference
Open label dose opt Clinical Global Impressions: Impairment and Severity (CGI I/S) | every visit (every 1-2 weeks over max of 12 weeks)
  completed at every visit ; 1 item each for impairment and severity on 1 to 7 likert; higher numbers mean more severity and less improvement; will examine change over time with med
Open label dose opt: Teacher Rated Inattention/Overactivity with Aggression (IOWA) | every visit (every 1-2 weeks over max of 12 weeks)
  completed every visit in this phase to measure change in ADHD symptoms at school; 10 items rated 0-4 with range from 0 to 40 and higher scores = more symptoms; will examine change over time with med
Open label dose opt: Guardian Rated Impairment Rated Scale (IRS) | every visit (every 1-2 weeks over max of 12 weeks)
  completed at every visit; 7 items covering 7 different domains; rated 0-6 with higher scores = more impairment; no total score; will examine change over time with med
Open label dose opt: Pittsburgh Side Effect Rating Scale (PSERS) | every visit (every 1-2 weeks over max of 12 weeks)
  completed by guardians at every visit; 11 items rated 0-4 (range 0-44) with greater side effect severity = higher scores; will examine change over time with med
Open label dose opt affective reactivity index clinician interview (CARI) | baseline (visit 1) and endpoint of this phase (max of 6 visits); each visit is spaced 1-2 weeks part so max time between measures would be 12 weeks
  completed by clinician interview of guardian ; covers 11 domains of irritability with total score 0 to 100 and higher scores representing more problems; will examine change over time with med
rct phase: affective reactivity index clinician interview (CARI) | completed weekly for two weeks
  completed by clinician interview of guardian ; covers 11 domains of irritability with total score 0 to 100 and higher scores representing more problems; will examine mean drug placebo difference
Open label dose opt: Disruptive Behavior Disorder Rating Scale (DBDRS) guardians | baseline (visit 1) and endpoint of this phase (max of 6 visits); each visit is spaced 1-2 weeks part so max time between measures would be 12 weeks
  completed by guardians at first and last visit to measure change in oppositional behaviors and other conduct problems; 45 items rated 0-3 with higher scores=more symptoms (range 0-135); will examine change over time with med
Open label dose opt: Disruptive Behavior Disorder Rating Scale (DBDRS) teachers | baseline (visit 1) and endpoint of this phase (max of 6 visits); each visit is spaced 1-2 weeks part so max time between measures would be 12 weeks
  completed by teachers at first and last visit to measure change in oppositional behaviors and other conduct problems; 45 items rated 0-3 with higher scores=more symptoms (range 0-135); will examine change over time with med
Open label dose opt: teacher rated impairment rating scale (IRS) | baseline (visit 1) and endpoint of this phase (max of 6 visits); each visit is spaced 1-2 weeks part so max time between measures would be 12 weeks
  measures student functioning at school; 7 items covering 7 different domains; rated 0-6 with higher scores = more impairment; no total score; will examine change over time with med
RCT Phase: Inattention/Overactivity with Aggression 5 item abridged EMA survey (IOWA) | 7 days on med and for 7 days on placebo for 14 days of data collection
  given by EMA to guardians daily for the 14 days of this phase; 5 items rated 0-4 with higher scores = worse symptoms (range 0-20); will examine drug placebo difference
RCT phase: Retrospective modified overt aggression scale (RMOAS) guardians | weekly for two weeks
  full version of RMOAS completed once per week by guardians; 12 items with first 4 items having 3 item likert and next 12 having 14 item likert; weighted score 0-20 for first 4 items measuring verbal incidents, 0-120 for next 4 items measuring incidents towards others and 0 to 60 for final set of 4 items measuring incidents to property for total range of 0 to 200 with higher scores meaning more aggressive behaviors; will examine drug placebo difference
RCT phase: Guardian rated Impairment Rating Scale (IRS) | weekly for two weeks
  to measure home impairment; 7 items covering 7 different domains; rated 0-6 with higher scores = more impairment; no total score; will examine drug placebo difference
RCT phase: Teacher rated Impairment Rating Scale (IRS) | weekly for two weeks
  to measure school impairment; 7 items covering 7 different domains; rated 0-6 with higher scores = more impairment; no total score; will examine drug placebo difference
RCT phase: Guardian rated Pittsburgh Side Effect Rating Scale (PSERS) | weekly for two weeks
  to measure medication tolerability; completed by guardians at every visit; 11 items rated 0-4 (range 0-44) with greater side effect severity = higher scores; will examine drug placebo difference
RCT phase: Teacher rated Affective reactivity Index (ARI) | weekly for two weeks
  range is 0-12 with higher scores representing more irritability; will examine drug placebo differnce
RCT phase: Teacher rated Retrospective modified overt aggression scale (RMOAS) | weekly for two weeks
  scale given weekly; 12 items with first 4 items having 3 item likert and next 12 having 14 item likert; weighted score 0-20 for first 4 items measuring verbal incidents, 0-120 for next 4 items measuring incidents towards others and 0 to 60 for final set of 4 items measuring incidents to property for total range of 0 to 200 with higher scores meaning more aggressive behaviors ; will examine drug placebo difference
Rct Phase: Teacher rated Inattention/Overactivity with Aggression (IOWA) | weekly for two weeks
  measures ADHD symptoms; 10 items rated 0 to 4 (0-40) with higher scores = more symptoms; will examine drug placebo difference
Reward positivity ERP | once per week RCT phase for total of two weeks
  measures response to reward feedback; will examine difference score between medication and placebo on winning quesses to see if it correlates with drug placebo difference score for ARI and RMOAS from this phase; measured in microvolts- no defined range
Switch Positivity ERP | once per week RCT phase for total of two weeks
  measures set shifting; will examine difference score between medication and placebo to see if it correlates with drug placebo difference score for ARI and RMOAS from this phase; measured in microvolts- no defined range
P3b ERP | once per week RCT phase for total of two weeks
  measured attentional allocation; will examine difference score between medication and placebo for P3b amplitude change during frustration vs non frustration blocks to see if it correlates with drug placebo difference score for ARI and RMOAS from this phase; measured in microvolts- no defined range

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Health Dept of Psychiatry, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified results for RACDS-25, DSM Crosscutting measure for youth (guardian completed) ARI, RMOAS, DBD-RS. IOWA, ADHDRS, PSERS, CGI, IRS, EEG data
Supporting Information: Study Protocol, SAP
Time Frame: consistent with policies for NIMH Data archive, dependent on notice of award date
Access Criteria: as per policies of the NIMH Data archive
URL: https://nda.nih.gov/